CLINICAL TRIAL: NCT06210698
Title: Angioedema Biomarker Research Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Foundation For Rare Disease Research (Other)
Collaborators: Institute for Asthma & Allergy (Unknown); Virant Diagnostics, Inc. (Unknown); MedBio Reference Laboratories, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: Virant-A001
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Angioedema; Angioedemas, Hereditary; Urticaria; Mastocytosis; ACE Inhibitor-Induced Angioedema; C1 Inhibitor Deficiency; Systemic Mastocytoses; Indolent Systemic Mastocytosis
Keywords: angioedema; c1-inhibitor deficiency; C1-inhibitor dysfunction; hereditary angioedema; HAE; ACE Inhibitor-induced angioedema; serum tryptase; mastocytosis; systemic mastocytosis; indolent systemic mastocytosis
MeSH Terms: conditions — Angioedema; Angioedemas, Hereditary; Urticaria; Mastocytosis; Mastocytosis, Systemic | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Plasma, Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent Angioedema: Broad definition: Angioedema due to urticaria (histaminergic/mast-cell) or non-urticarial (non-histaminergic) etiology Narrow definition: non-urticarial angioedema - distinguishing between C1-Inhibitor deficiency/dysfunction, and Angioedema with normal levels of C1-Inhibitor.
  Interventions: Diagnostic Test: Venipuncture
- Healthy Subjects: Broad definition: No medical history of angioedema of any kind, including urticaria (histaminergic) or drug-induced angioedema (e.g. ACE-Inhibitor angioedema)
  Interventions: Diagnostic Test: Venipuncture

INTERVENTIONS:
Diagnostic Test: Venipuncture — venipuncture

SUMMARY:
This clinical trial aims to evaluate and compare novel and commercially available diagnostic assays through blood tests for the differential diagnosis and comprehensive assessment of patients experiencing recurrent angioedema attacks, including both urticarial and non-urticarial angioedema. The primary objective is to assess the efficiency of novel diagnostic assays, both individually and in combination, in comparison to currently available commercial tests. The ultimate goal is to establish the feasibility of developing an affordable and accurate laboratory test capable of diagnosing the diverse etiological manifestations of angioedema.

DETAILED DESCRIPTION:
Purpose: The purpose of this prospective non-interventional non-randomized diagnostic study is to first identify patients with recurrent angioedema attacks, then collect their blood samples (venipuncture) and ultimately send the samples to specialized laboratories to perform multiple diagnostic assays, novel and traditional, that can distinguish the various forms of angioedema (urticaria and non-urticarial symptoms and signs), and healthy subjects.

Methods and Materials: Blood specimen collection from a total of 300 patients with recurrent angioedema attacks, and 300 healthy volunteers without a history of angioedema attacks. Laboratory testing will include assays on multiple platforms. Complement testing via immunoassay and biochemistry techniques. Flow Cytometry using multiple markers. Mass Spectrometry that includes bradykinin metabolite and histamine detection. Molecular Genetics include Sanger sequencing, Next Generation Sequencing (NGS), and digital PCR.

Patient population: Study participants to be screened who have a history of recurrent angioedema incidents as well as a population of healthy subjects. A medical history will be documented after obtaining informed patient consent to enter into the clinical trial. Each enrolled participant will have blood collected as whole blood, plasma and serum via venipuncture.

Eligibility criteria (inclusion) for sample collection (angioedema subject):

* Understand and sign the informed consent form before starting any study procedure.
* Adult or Child: aged 12 years of age or older (consent must be signed by a single parent or legal guardian).
* Angioedema symptoms and signs by medical history, or previous laboratory diagnostic testing, or genetically proven cases (e.g. SERPING1 or other mutation). Patients can be on active medication for the treatment and prophylaxis of angioedema. Angioedema cases must be verified by a clinician from IAA.
* Able to perform and endure safely the collection of peripheral blood samples (venipuncture), or optionally agree to have additional testing via a skin punch biopsy.

Eligibility criteria (inclusion) for sample collection (for healthy participant/subject):

* Understand and sign the informed consent form before starting any study procedure.
* Adult or Child: aged 12 years of age or older (consent must be signed by a single parent or legal guardian).
* No history of any angioedema symptoms and signs, previous laboratory diagnostic testing, or genetically proven cases.
* Able to perform and endure safely the collection of peripheral blood samples (venipuncture), or optionally agree to have additional testing via a skin punch biopsy.
* Not on ACE inhibitors and if on blood pressure medication, to indicate the drug(s).

Exclusion Criteria (for all participants):

* Minor: 11 years of age or younger.
* Cannot read or understand the informed consent form and instructions.
* Unable to perform the peripheral blood sample collection.
* Taking medications contraindicated for testing.
* History of excessive bleeding after phlebotomy, e.g. Hemophilia.
* Contraindication due to other health-related issues.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign the informed consent form before starting any study procedure.
* Adult or Child: aged 12 years of age or older (consent must be signed by a single parent or legal guardian).
* Angioedema symptoms and signs by medical history, or previous laboratory diagnostic testing, or genetically proven cases (e.g. SERPING1 or other mutation). Patients can be on active medication for the treatment and prophylaxis of angioedema. Angioedema cases must be verified by a clinician from IAA.
* Able to perform and endure safely the collection of peripheral blood samples (venipuncture), or optionally agree to have additional testing via a skin punch biopsy.

Exclusion Criteria:

* Minor: 11 years of age or younger.
* Cannot read or understand the informed consent form and instructions.
* Unable to perform the peripheral blood sample collection.
* Taking medications contraindicated for testing.
* History of excessive bleeding after phlebotomy, e.g. Hemophilia.
* Contraindication due to other health-related issues.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The collection of medical history and peripheral blood (venipuncture) to perform multiple diagnostic assays from patients experiencing recurrent angioedema attacks, including both urticarial and non-urticarial angioedema. Healthy volunteers will not have a medical history of angioedema.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Novel versus traditional diagnostic blood test for angioedema | 2 years
  Determining whether novel test methods can be more efficient than currently available or traditional laboratory test for angioedema diagnosis

SECONDARY OUTCOMES:
Genetic analysis of angioedema versus non-angioedema affected populations | 2 years
  Genetic testing that include know angioedema mutations, such as SERPING1
Development of novel Bradykinin biomarkers | 2 years
  Mass Spectrometry analysis of plasma for bradykinin metabolites
Immunoassay laboratory developed tests for angioedema | 2 years
  development of novel immunoassay biomarkers, such as the detection of cleaved HMWK
Lymphocyte profile studies | 2 years
  Determine whether the immune system has a role in angioedema attacks

CONTACTS AND LOCATIONS:
Overall Officials: Lili Wan, PhD, Study Director — Institute for Asthma & Allergy

IPD SHARING:
Plan to Share IPD: Yes
The analyzed data will be published in a peer-reviewed journal and preliminary results published on clinicaltrials.gov website
Supporting Information: Study Protocol, CSR
Time Frame: 2 years